CLINICAL TRIAL: NCT05336604
Title: Epidémiologie et Conditions de Vide liées au Covid-19 STUDY OF THE COVID-19 (SARS-CoV-2) EPIDEMIC AND SOCIO-ECONOMIC LIVING
Brief Title: STUDY OF THE COVID-19 EPIDEMIC AND SOCIO-ECONOMIC LIVING CONDITIONS IN FRANCE
Acronym: EpiCov
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-25; 2020-A01191-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: General Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Home blood self-sample on dried blood spot (DBS) to perform COVID-19 serology Serological tests was based on a home self-capillarous blood samples collected by the participants, from a finger prick dried blood spot 903 Whatman paper (DBS) kits, subsequently analyzed in a centralized virology laboratory. At the biobank, DBS cards were punched using a PantheraTM machine (PerkinElmer). The tubes were sent to the virology laboratory (Unité des virus Emergents, Inserm/IRD, Marseille, France), in order to detect IgG antibodies against the spike protein (Euroimmun ELISA-S), and neutralizing antibodies for non-negative ELISA-S.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population, aged 15 years or more, living in France: Population-based ohort of general population, aged 15 years or more, living in France in May 2020, selected at random from national administrative sample frame

SUMMARY:
EpiCov is a population-based cohort which aims to provide national and regional estimates of seroprevalence of SARS-CoV-2 infection and analyse relations between living conditions and the dynamics of the epidemic in France. The study population is a random sample of individuals aged 15 years and older, excluding people living in residences for the elderly and living in jail. The participants are recruited from the French national tax register and is representative of the population living in France. Home self-samples on Dried Blood Spots (DBS) for IgG and neutralizing antibodies detection were offered to a random national sub-sample of 12,114 in the 1st round of the EPICOV survey (May 2020) and to all respondents in the 2nd round (November 2020), including also serological testing for all members (≥ 6 years old) of household for 20% of index participants. A third round was perfomed in June-July 2021, without serological measurements. Overall, 134,391 participants have been enrolled in first-round (May 2020). Among them, 107 759 participated to the second round (November 2020) and 85 074 in third round (June 2021). The next wave is expected in March-april 2022.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 15 years or older
* living on January 1, 2020, in mainland France or one of three overseas departments (Martinique, Guadeloupe and Réunion Island).

Exclusion Criteria:

* individuals living in prisons at the time of the study
* people living in residential institutions for dependent elderly persons, as caregivers were not available during the epidemic period to help them with internet access or phone calls.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population-based sample based on a national random probability sample from the administrative sample frame: all individuals aged 15 years or older on January 1, 2020, living in mainland France or one of three overseas departments (Martinique, Guadeloupe and Réunion Island). Due to the poor quality of the sampling frame, poor internet access and the use of multiple languages, two other overseas departments, French Guiana and Mayotte, were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 134391 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Changes in COVID-19 Seroprevalence over time | Inclusion, 6 months, 14 months, 28 months
  Proportion of the individuals tested with an Euroimmun ELISA-S ratio >1.1 (ELISA S+), from home self-sampling on capillarous blood sampled.
  Serological tests was based on a capillarous blood samples collected by the participants themselves, at home, from a finger prick dried blood spot 903 Whatman paper (DBS) kits, which was subsequently analyzed in a centralized virology laboratory. The sample kits were delivered by express mail to each participant who had sent their samples by mail to the EpiCov biobank. At the biobank, DBS cards were punched from the spots on the Whatman paper, using a PantheraTM machine (PerkinElmer). The tubes were sent to the virology laboratory (Unité des virus Emergents, Inserm/IRD, Marseille, France), in order to detect IgG antibodies against the spike protein (Euroimmun ELISA-S), and neutralizing antibodies for non-negative ELISA-S.
Changes in living condition | Inclusion, 6 months, 14 months, 28 months
  Questions relating to living conditions were included: socioeconomic characteristics, size and nature of the habitation, number of people in the household, working condition, childcare, home-schooling, inter-partner relationships within the household
Changes in health condition | Inclusion, 6 months, 14 months, 28 months
  Health status was described through general and specific questions regarding self-perceived health, symptoms potentially linked to COVID-19, mental health, and access to healthcare, whether or not linked to COVID-19.
COVID-19 IgG antibodies median | 28 months
  Median of Euroimmun ELISA-S IgG, from home self-sampling on capillarous blood sampled.

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm U1018, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Yes
The EpiCov data is available for research purpose, 9 months after overall completion of one round. Access to anonymized individual data may be available before the planned period of open access : specific project has to be presented to the EpiCov exploitation committee : if accepted, it needs approval of ethics and reglementary Committee for researchers who meet the criteria for access to data.
  The first round, and will be available by March 2022 concerning the second round for research purpose on CASD (https://www.casd.eu/), after submission to approval of French Ethics and Regulatory Committee procedure (Comité du Secret Statistique, CESREES and CNIL).
Supporting Information: Study Protocol, ICF
Time Frame: The first round is currently available and the second rond will be available by March 2022
Access Criteria: Access for research purpose of first and second round on CASD (https://www.casd.eu/) is given after submission to approval of French Ethics and Regulatory Committee procedure (Comité du Secret Statistique, CESREES and CNIL).
  Access to data for subsequent rounds may be available before the planned period of open access : specific project has to be presented to the EpiCov exploitation committee : if accepted, it needs approval of ethics and reglementary Committee for researchers who meet the criteria for access to data.